CLINICAL TRIAL: NCT04041453
Title: Prospective, Parallel-group, Open-label Randomized Controlled Trial of Four Treatment Regimes for Trichuriasis in Pediatric Patients
Brief Title: Albendazole Plus High Dose Ivermectin for Trichuriasis in Pediatric Patients
Acronym: HI4T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alejandro Krolewiecki (Other)
Collaborators: Brock University (Other); Universidad Nacional del Centro de la Provincia de Buenos Aires (Other); Universidad Nacional Autonoma de Honduras (Other)
Responsible Party: Sponsor-Investigator, Alejandro Krolewiecki, Investigador CIC CONICET, Universidad Nacional de Salta
Organization: Universidad Nacional de Salta (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-2019
Record Dates: First submitted 2019-07-22; First posted 2019-08-01 (Actual); Results first posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Trichuris Infection; Helminthiasis
Keywords: TRICHURIS; STH; IVERMECTIN; ALBENDAZOLE
MeSH Terms: conditions — Trichuriasis; Helminthiasis | interventions — Ivermectin; Albendazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Albendazole 400mg (Active Comparator): Albendazole 400mg in single dose
  Interventions: Drug: Albendazole
- Albendazole/Ivermectin (Experimental): Combination of albendazole 400mg + ivermectin 600mcg/kg in single dose.
  Interventions: Drug: Ivermectin; Drug: Albendazole
- Albendazole 400mg x 3 (Experimental): Albendazole 400mg/day for 3 consecutive days
  Interventions: Drug: Albendazole
- Albendazole/Ivermectin x 3 (Experimental): Combination of albendazole 400mg/day + ivermectin 600mcg/kg/day for 3 consecutive days
  Interventions: Drug: Ivermectin; Drug: Albendazole

INTERVENTIONS:
Drug: Ivermectin — Ivermectin at 600mcg/kg in addition to albendazole will be provided for 1 or 3 days.
  Arms: Albendazole/Ivermectin; Albendazole/Ivermectin x 3
Drug: Albendazole — Albendazole will be provided as an active control or in experimental arms for 1 or 3 days with ivermectin.

SUMMARY:
There are four species of intestinal worms collectively known as soil-transmitted helminthiasis (STH): Ancylostoma duodenale and Necator americanus (hookworms), Ascaris lumbricoides (roundworms), and Trichuris trichiura (whipworms). These parasites affect over two billion people and contribute to significant morbidity and disability, especially in high risk groups, for example children, agricultural workers and pregnant women. In children, STH are associated with impaired nutritional status evidenced by stunting, thinness and underweight.

As is the case in most Latin America, STH are a public health problem in Honduras. The World Health Organization (WHO) informs that more than 2.5 million children (under 15 years of age) in the country are at risk of infection. To control these infections Honduras has established a national deworming program that operates since 2001 but despite these efforts, the prevalence of STH infections remains unacceptably high. This is especially true in rural communities where prevalence can be as high as 70% of the children population.

Ivermectin (IVM) in combination with albendazole (ALB) has demonstrated the capacity to improve efficacy compared to any of these drugs in monotherapy; the efficacy is however, still inadequate in terms of cure rate, although egg reduction rates are significant.

The purpose of the current trial is to assess the safety and efficacy of 3 experimental regimens for the treatment of infections by Trichuris trichiura in children in comparison with the current standard of practice in Mass Drug Administration (MDA) campaigns. The experimental regimens will explore the effect of multiple day regimens and high dose ivermectin.

Treatment arms:

* Group 1: single dose of ALB 400 mg. (active control arm). N:39
* Group 2: single dose ALB 400mg + IVM 600µg/Kg. N: 57
* Group 3: daily dose ALB 400mg for 3 consecutive days. N:24
* Group 4: daily dose ALB 400mg + IVM 600µg for 3 consecutive days. N:57

Total Study Population: 177

ELIGIBILITY:
Inclusion Criteria:

* Infection with T. trichiura by Kato Katz.
* Body weight >15kg.
* Accepts participation

Exclusion Criteria:

* Albendazole and/or mebendazol treatment in the previous 3 months.
* Allergy to the study drugs
* Acute medical conditions
* Clinical trial participation in the previous 3 months.
* Pregnancy.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro J Krolewiecki, MD, PhD, Study Director — IIET - Universidad Nacional de Salta
Locations (2):
- IIET, Orán, Salta Province, Argentina
- Universidad Autónoma de Honduras, Tegucigalpa, Honduras

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Analytic Code
Time Frame: After study data analysis completion, with submission for publication to a peer review journal..
Access Criteria: Database will be made available through a publication.

REFERENCES:
- [Derived] Matamoros G, Sanchez A, Cimino R, Krolewiecki A, Mejia R. A comparison of the diagnostic capability of Kato-Katz and real-time PCR for the assessment of treatment efficacy of ivermectin and albendazole combination against T. trichiura infections. PLoS Negl Trop Dis. 2024 Nov 19;18(11):e0012677. doi: 10.1371/journal.pntd.0012677. eCollection 2024 Nov. PMID 39561184
- [Derived] Matamoros G, Sanchez A, Gabrie JA, Juarez M, Ceballos L, Escalada A, Rodriguez C, Marti-Soler H, Rueda MM, Canales M, Lanusse C, Cajal P, Alvarez L, Cimino RO, Krolewiecki A. Efficacy and Safety of Albendazole and High-Dose Ivermectin Coadministration in School-Aged Children Infected With Trichuris trichiura in Honduras: A Randomized Controlled Trial. Clin Infect Dis. 2021 Oct 5;73(7):1203-1210. doi: 10.1093/cid/ciab365. PMID 33906234

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Albendazole 400mg | Albendazole/Ivermectin | Albendazole 400mg x 3 | Albendazole/Ivermectin x 3
Started | 38 | 57 | 23 | 58
Safety Population | 38 | 56 | 23 | 58
Completed | 24 | 35 | 18 | 40
Not Completed | 14 | 22 | 5 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albendazole 400mg | Albendazole/Ivermectin | Albendazole 400mg x 3 | Albendazole/Ivermectin x 3 | Total
Number analyzed (Participants) | 38 | 57 | 23 | 58 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (2.6) | 8.0 (2.2) | 8.5 (2.0) | 8.0 (2.2) | 8.2 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 13 | 30 | 86
  Male | 19 | 33 | 10 | 28 | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate
Description: Number of individuals cured from Trichuris trichiura infection using the duplicate Kato Katz laboratory method on a single sample of fresh stools as the measurement tool. Cure rate is defined as the absence of Trichuris trichiura eggs in post-treatment samples.
Time Frame: 21 days
Population: The follow-up visit for efficacy assessment on Day 21 post-drug administration was not conducted in 52 subjects due to the outbreak of COVID-19 pandemic in Honduras which precluded completion of study visits in March 2020.
  Additional 7 subjects did not complete the study: 1 did not take the study medication, and 6 subjects were lost to follow up.
Measure: Count of Participants; unit: Participants
Groups:
- Albendazole 400mg x3: Albendazole 400mg/day for 3 consecutive days.
Arm/Group | Albendazole 400mg | Albendazole/Ivermectin | Albendazole 400mg x3 | Albendazole/Ivermectin x 3
Number analyzed (Participants) | 24 | 35 | 18 | 40
Participants | 1 | 31 | 6 | 40

2. Secondary Outcome: Egg Change Rate
Description: Calculation details: 100 x (1 - arithmetic mean fecal egg count post-intervention / arithmetic mean fecal egg count pre-intervention) Egg change rate was calculated across all participants, as described in reference: Levecke B et al., PLoS Negl Trop Dis. 2014;8(10).
Time Frame: 21 days
Population: as for outcome 1
Measure: Number; unit: Percent change
Groups:
- Albendazole/Ivermectin: Albendazole 400mg + ivermectin 600mcg/kg in single dose.
- Albendazole x 3: Albendazole 400mg/day for 3 consecutive days.
Arm/Group | Albendazole 400mg | Albendazole/Ivermectin | Albendazole x 3 | Albendazole/Ivermectin x 3
Number analyzed (Participants) | 24 | 35 | 18 | 40
Percent change | 50 | 97 | 72 | 100

3. Secondary Outcome: Beta Tubulin Resistance
Description: Measurement of the incidence of mutations of tubulin in Trichuris trichiura eggs collected pre and post treatment using molecular biology techniques.
  This data is not available yet due to the COVID-19 pandemic, but the data will be available and reported in the future. Anticipated reporting date for this outcome measure is estimated by 2021 and will be confirmed once the pandemic is over.
Time Frame: 21days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected since the subject's enrollment until end of study participation (Day 21).
Groups:
- Albendazole 400mg x3: Albendazole 400mg/day in 3 consecutive days
- Albendazole/Ivermectin x 3: Combination of albendazole 400mg/day + ivermectin 600mcg/kg/day in 3 consecutive days
Arm/Group | Albendazole 400mg | Albendazole/Ivermectin | Albendazole 400mg x3 | Albendazole/Ivermectin x 3
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/56 | 0/23 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/56 | 0/23 | 0/58
Other Adverse Events (participants affected / at risk) | 0/38 | 10/56 | 7/23 | 10/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albendazole 400mg (N=38) | Albendazole/Ivermectin (N=56) | Albendazole 400mg x3 (N=23) | Albendazole/Ivermectin x 3 (N=58)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (General disorders) | 0 (0) | 5 (5) | 2 (2) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT04041453/Prot_SAP_000.pdf